CLINICAL TRIAL: NCT00913263
Title: An Open, Single and Multiple Dose, Efficacy and Safety Proof of Principle Study of Liproca Depot, a Controlled Release Formulation of 2-hydroxyflutamide, Injected Into the Prostate in Patients With Localized Prostate Cancer
Brief Title: An Efficacy and Safety Study With Licroca Depot, a Controlled Release Product, Injected Into the Prostate
Acronym: 2-HOF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lidds AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPC-002; 2009-010079-25 (EudraCT Number)
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — hydroxyflutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2-Hydroxyflutamide (Experimental): Single injection of 2-Hydroxyflutamide (2-8mL ready-made paste)in one prostate lobe
  Interventions: Drug: 2-hydroxyflutamide (2-HOF) [Liproca Depot]; Drug: 2-Hydroxyflutamide

INTERVENTIONS:
Drug: 2-hydroxyflutamide (2-HOF) [Liproca Depot] — Ready made paste including 600 mg 2-HOF for injection as a single dose
  Other Names: Liproca Depot
Drug: 2-Hydroxyflutamide — The Product consists of two sterile components, one aqueous liquid and a dry powder, containing the active drug 2-Hydroxyflutamide (2-HOF. The two components were mixed under aceptic conditions to a paste prior to administration.
  Other Names: Liproca Depot

SUMMARY:
The primary objective was to evaluate efficacy of a single dose of Liproca Depot in patients with localized prostate cancer. Primary efficacy variable was the proportion of patients showing PSA nadir. 24 Caucasian men, with a mean age at inclusion of 68.4 years, with localized prostate cancer were injected once with a ready made paste including 600 mg 2-hydroxyflutamide (Liproca Depot) into the site of the prostate where the tumour was localized. The patient was monitored for prostate-specific antigen (PSA) for maximum 6 months or to progression within this time period. The primary endpoint showed interesting results with high success rate (83%), i.e. proportion of patients (Responders) that reached plasma PSA nadir.

DETAILED DESCRIPTION:
Patients with localized prostate cancer were followed to progression or maximum 24 weeks after a single injection in one lobe of 2-8 mL ready-made paste (corresponding to 400-1600 mg 2-Hydroxyflutamid). Progression was defined as an increase in PSA by > 25% over baseline or on-treatment nadir.Among the 24 patients the primary endpoint, plasma PSA nadir, was reached by 20 patients (Responders). Efficacy was measured primarily as PSA nadir, and secondly as time to PSA nadir and prostate volume change. Safety was monitored throughout the whole study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45years
2. Histologically confirmed localized prostate cancer (T1-T2), predominantly in one side of the peripheral zone, verified by biopsy.
3. PSA value < 20 ng/ml within 6 weeks before enrolment.
4. Gleason score ≤ 3+4 at diagnostic biopsy
5. Adequate renal function: Creatinine < 1.5 times upper limit of normal.
6. Adequate hepatic function: ASAT, ALAT and ALP < 1.5 times upper limit of normal.
7. Negative dipstick for bacturia.
8. Patient must have ability to cope with the study procedures and to return to scheduled visits including follow up visit.

Exclusion Criteria:

1. Previous or ongoing hormone therapy for prostate cancer.
2. Ongoing or previous therapy (within3 month) of finasteride or dutasteride.
3. Ongoing or previous invasive therapy for benign prostate hyperplasia (TURP, TUMT).
4. Symptoms or signs of acute prostatitis.
5. Symptoms or signs of ulceric proctitis
6. Severe micturation symptoms (I-PSS >17)
7. Concomitant systemic treatment with corticosteroids, or immunomodulating agents.
8. Known immunosuppressive disease (e.g. HIV, insulin dependent diabetes).
9. Simultaneous participation in any other study involving not market authorized drugs or having participated in a study within the last 12 months prior to start of study treatment.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo Tammela, Professor, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the pool of patients with prostate cancer (T1-T2) available at the clinic. They were informed about the study by the Investigator
Pre-assignment Details: There was only one Group assignment for the study. The patients (men with histologically confirmed localized prostate cancer, verifyed by biopsy), aged ≥ 45 years, with PSA value <20ng/mL, within 6 weeks before enrollment, and and Gleason score <3+4 at diagnostic biopsy.
Groups:
- Hydroxyflutamide (2-HOF): Men with histologically confirmed localized prostate cancer (T1-T2) predominantly in one side of the periferal zone, verified by biopsy. Age ≥ 45 years.
Period: Overall Study
Arm/Group | Hydroxyflutamide (2-HOF)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Men with histologically confirmed localized prostate cancer (T1-T2) predominantly in one side of the periferal zone, verified by biopsy. Age ≥ 45 years.
Arm/Group | Group 1
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Region of Enrollment [Number; unit: participants]
  Finland | 24

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Showing PSA Nadir
Description: Plasma PSA nadir is the lowest PSA reading achieved after any treatment for prostate cancer. The patients were observed once every 4th week during the study period.
Time Frame: Measured every 4th week until progression or maximum 6 months.
Population: All patients who received the single dose of Liproca® Depot and had a baseline plasma PSA measurement, and at least one PSA measurement after the baseline measurement, were included in the efficacy analysis.
  Study population safety All patients who received at least one dose of Liproca® Depot were included in the safety analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients with PSA nadir
Groups:
- Part I: Patients () 24 patients) in Part I have been injected with Liproca Depot once. Patients in Part II (9 patients)have been injected twice with Liproca Depot. The second injection was after progression in Part I.
Arm/Group | Part I
Number analyzed (Participants) | 24
percentage of patients with PSA nadir | 83 [63 to 95]

2. Secondary Outcome: Number of Patients Reporting Adverse Events Caused by the Study Treatment
Description: * Adverse events caused by the study treatment
  * Abnormal, clinically relevant, laboratory parameters
  * Voiding symptoms
  * Vital Signs
  * Quality of Life
Time Frame: Measured every 4th week till progression or maximum 6 months
Population: All patients who received the single dose of Liproca® Depot and had a baseline plasma PSA measurement, and at least one PSA measurement after the baseline measurement, should be included in the efficacy analysis.
  Study population safety All patients who received at least one dose of Liproca® Depot should be included in the safety analysis.
Measure: Number; unit: Patients reporting study related AE
Groups:
- Group 1: 24 patients (Part I of the study) have been injected with Liproca Depot once.
Arm/Group | Group 1
Number analyzed (Participants) | 24
Patients reporting study related AE | 12

3. Secondary Outcome: Percent Change in Prostate Volume From Baseline to Nadir.
Description: Prostate volume was measured at each visit to capture nadir and compared to baseline for all patients. Decrease in prostate volume is reported as percent change from baseline.
Time Frame: Measured every 4th week until progression or maximum 6 months.
Measure: Median (Standard Deviation); unit: percent change
Groups:
- Part I: Patients (24 patients) in Part I have been injected with Liproca Depot once.
Arm/Group | Part I
Number analyzed (Participants) | 24
percent change | 14 (9.6)

4. Secondary Outcome: Time to PSA Nadir
Description: Time frame was from baseline to day of PSA nadir.
Time Frame: Measured every 4th week until progression or maximum 6 moths.
Measure: Number (95% Confidence Interval); unit: Number of days from baseline to PSA nadi
Groups:
- Part I: Patients () 24 patients) in Part I have been injected with Liproca Depot once.
Arm/Group | Part I
Number analyzed (Participants) | 24
Number of days from baseline to PSA nadi | 77 [32 to 126]

5. Secondary Outcome: Percent Change in Prostate Volume From Baseline to Final Visit
Description: Prostate volume was captured at each visit and percent change from baseline to final visit was measured. Final visit was either day of progression or after 6 months. Prostate volume decrease is reported in percent change from baseline
Time Frame: Measured every 4th week until progresion or maximum 6 months.
Measure: Median (Standard Deviation); unit: percentage change
Arm/Group | Part I
Number analyzed (Participants) | 24
percentage change | 7 (11)

6. Secondary Outcome: Number of Days to Prostate Volume Nadir.
Description: Number of Days from day of injection to prostate volume nadir.
Time Frame: Measured every 4th week until progression or maximum 6 months.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Part 1: Patients (24 patients) have been injected with Liproca depot once
Arm/Group | Part 1
Number analyzed (Participants) | 24
Days | 112 [21 to 184]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=24)
Prostate infection (Infections and infestations) | 1 (1) — The event was caused by the injectiontechnique
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=24)
dysuria, haematuria (Renal and urinary disorders) | 12 (16)

LIMITATIONS AND CAVEATS:
There were no limitations of the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No